CLINICAL TRIAL: NCT03347032
Title: Remote Ischemic Preconditioning for Renal Protection in Patients Undergoing Transcatheter Aortic Valve Interventions
Brief Title: Remote Ischemic Preconditioning for Renal Protection in TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Brittany Fuller, MD, Co-Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIPC TAVI
Record Dates: First submitted 2017-11-08; First posted 2017-11-20 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Aortic Valve Stenosis; Renal Insufficiency; Contrast-induced Nephropathy
MeSH Terms: conditions — Aortic Valve Stenosis; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will undergo remote ischemic preconditioning with serial inflations of the blood pressure cuff to 200 mmHg followed by deflation for reperfusion for a period of 5 minutes each for a total of 4 cycles.
  Interventions: Procedure: Remote ischemic preconditioning
- Control (Sham Comparator): This group will undergo serial inflations of the blood pressure cuff to 40 mmHg followed by deflation for a period of 5 minutes each for a total of 4 cycles.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Serial inflations and deflations as detailed in the arm/group descriptions
  Arms: Intervention
Procedure: Control — Serial inflations and deflations as detailed in the arm/group descriptions
  Arms: Control

SUMMARY:
Severe aortic stenosis remains a major cause of morbidity and mortality of the elderly affecting approximately 3% of elderly patients with an increasing number of patients undergoing transcatheter aortic valve interventions. As part of pre-procedural planning these patients undergo CT scans and receive contrast during the procedure. These patients often have baseline renal insufficiency and are high risk of contrast induced nephropathy despite pre-hydration techniques. The purpose of this study is to evaluate the efficacy of this simple and safe procedure in preventing renal injury in this particular population.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged 18 or older presenting with moderate to severe aortic stenosis for a trans-catheter aortic valve intervention

Exclusion Criteria:

* Patients in cardiogenic shock defined as requiring circulatory or hemodynamic support with a device, vasopressors or inotropes
* Systemic hypotension (systolic blood pressure < 90mmHg)
* Patients currently on hemodialysis
* Presence of an arteriovenous dialysis fistula or graft or lymphedema in either arm
* Patients enrolled in other active cardiovascular investigational studies
* Severe comorbidities with a life expectancy of less than 6 months
* Pregnant or lactating women
* Patients unable to provide consent
* Patients taking the medication glibenclamide for treatment of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Renal function as a measured by serum creatinine | 48-72 hours
  Assess the effects on post procedure renal injury. Lab work will be obtained in the form of a basic metabolic panel evaluating the creatinine level. A baseline basic metabolic panel will be obtained prior to scheduled procedure to evaluate baseline renal function and then 48-72 hours post procedure, the optimal time to see the effects of contrast induced nephropathy to evaluate the degree of acute kidney injury. The baseline and post procedure measurements of renal function will be compared between both arms of the study.

SECONDARY OUTCOMES:
Clinical Outcomes | 6 months
  The patient's electronic medical record will be reviewed at 6 months post procedure. The investigators will be assessing renal function at 6 months if a creatinine (lab) was ordered by the primary provider for any reason.
Clinical Outcomes | 6 months
  The investigators will be reviewing the medical records of participants for evidence of post procedure adverse events including death, MI, stroke and hospital readmission

CONTACTS AND LOCATIONS:
Overall Officials: William O'Neill, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States